CLINICAL TRIAL: NCT02837159
Title: Effectiveness of a Mobile Application for the Promotion of Healthy Lifestyle Habits in Patients With Colorectal Cancer: a Randomized Controlled Trial
Brief Title: A Mobile Aplication for the Promotion of Healthy Lifestyle Habits in Patients With Colorectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: removal of the Phd student due to not obtaining financing
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, Dra, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CO217
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; Health Life Style Habits; Health
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- mHealth application (Experimental): The assessment of the end points will be made at three moments: at baseline, at 8 weeks (at the end of the program) and at 12 months of follow-up. The intervention will consist in: 1)Feedback daily or weekly of physical exercise and diet through the application (notice) according to the records of diet and exercise and following recommendations of International Organizations 2) Participation in three sessions of seminars (1 hour each every 15 days) on habits of life healthy and cancer and the self-regulation through measurements performed by the application 3) Calls weekly to the patients of way individual to comment possible errors or doubts about the application, of 10 min of duration (8 calls).
  Interventions: Other: mHealth application
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: mHealth application — Dietary and physical activity recommendations trough a mobile application
  Arms: mHealth application

SUMMARY:
The purpose of this randomized study is to assess the efficacy of a mobile application for the promotion of healthy lifestyle habits (diet and exercise) in colorectal cancer survivors (CCR).

DETAILED DESCRIPTION:
Background: Among all types of cancer, colorectal cancer (CRC) is one of the most frequent, and Spain is among the countries with the highest incidence of CCR with a ratio of about 100,000 people. Fortunately the data of survival are very encouraging according to the National Cancer Institute, it is around 70% at 5 years when the cancer is regional and it could reaching up to 90% when it is more localized. During this survival, however, a high number of patients suffer physical and psychological sequelae that limited their quality of life.

This is why that, to try to minimize these effects, it is essential to try to instill healthy habits (food and physical exercise), since as it confirms the current literature, obesity is related to a lower survival and a greater presence of other diseases, and increased consumption of fruits and vegetables and physical activity practice improves the quality of life in survivors of CRC. However, changes in lifestyle are complicated to maintain long-term. In this sense, the technological development offers possibilities to try to resolve this lack of adherence in patients with cancer. However, the evidence highlights the need to improve knowledge about its applicability and efficacy in patients with this pathology betting on technologies more innovative.

Objective: The purpose of this randomized study is to assess the efficacy of a mobile application for the promotion of healthy lifestyle habits (diet and exercise) in CRC survivors. In a more specific way, analyze the effectiveness of the implementation to maintain healthy lifestyle habits in patients newly diagnosed with CRC through adherence to a healthy lifestyle (exercise and diet), as well as facilitate changes in clinical variables: body composition, quality of life, physical condition related to health (functional ability, strength and flexibility).

Methods: 54 patients will be recruited from the Virgen de las Nieves Hospital from Granada (Spain). Patients will be randomized in two groups: control and experimental group. The assessment of the end points will be made in IMUDS (Instituto Mixto Deporte y Salud) from Granada (Spain) at three moments: at baseline, at 8 weeks (at the end of the program) and at 12 months of follow-up. The intervention will consist in: 1)Feedback daily or weekly of physical exercise and diet through the application (notice) according to the records of diet and exercise and following recommendations of International Organizations 2) Participation in three sessions of seminars (1 hour each every 15 days) on habits of life healthy and cancer and the self-regulation through measurements performed by the application 3) Calls weekly to the patients of way individual to comment possible errors or doubts about the application, of 10 min of duration (8 calls). The control group will follow the usual indications of their oncologist and completion of the study will be offered access to the application.

Discussion: Health mobile applications (mobile health, mHealth) are potential tools to address the needs of cancer patients, because it enabling personalized interventions and the adherence to them. Previous studies have showed: 1) Are effective for weight loss in people with obesity or overweight. 2) You can count on are to promote a healthy lifestyle focused on the loss of weight in cancer patients. 3) Strategies based on self-regulation will not only improve the regulation of the exercise by the patient, but they also produce a greater adherence to the same. However, despite all these advances, are few them studies that have analyzed the efficiency of mobile applications as tool appropriate for foster the acquisition of habits of life healthy in cancer patients. Therefore are necessary studies that improve the adequacy of interventions to the needs of patients with CRC with support from technologies that show its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosed of colorectal cancer (estadio I-IIIa)
* Have finished the primary medical treatment.
* Have a body mass index > 25
* Have a level of physical activity < 3 METS
* Have access to a Smartphone

Exclusion Criteria:

* Physical effort Contraindication from their oncologist
* Anemia
* Presence of pathologies that make more difficult the practice of physical activity such as osteoarthritis.
* Inability to read
* Severe depression, physical deficits or cognitive
* Participation in any program or intervention for weight control

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2018-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | Participants will be followed over 12 months
  in kg/m2, will be assessed by conducting Dual-energy X-ray absorptiometry (DXA, discovery densitometer from HOLOGIC, QDR 4500W)

SECONDARY OUTCOMES:
Fat mass | Patients will be followed over 12 months
  Fat mass (%): will be evaluated by conducting Dual-energy X-ray absorptiometry (DXA, discovery densitometer from HOLOGIC, QDR 4500W)
Wait circunferemce | Patients will be followed over 12 months
  It will be measured with a plastic tape. Waist circumference was assessed midway between the lower rib margin and the top of the iliac crest (cm) at the end of normal breathing.
Hip circunferemce | Patients will be followed over 12 months
  It will be measured with a plastic tape. Hip circumference was measured at the level of the greater trochanter.
Expenditure energy | Patients will be followed over 12 months
  it will be assessed though FITBIT CHARGE HR bracelet in kcal/day.
Eating habits | Patients will be followed over 12 months
  through a record of 24-hour, recording the amount of macronutrients (carbohydrates, lipids, proteins), micronutrients (vitamins and minerals), fiber and energy density.
Cardiorespiratory fitness | Patients will be followed over 12 months
  the 6 minutes walking test will be used to measure the distance (m) that patients could walk in 6 minutes.
Isometric abdominal strength | Patients will be followed over 12 months
  it will be assessed with trunk curl test. Patient through a trunk curl has to keep an isometric position separating the inferior angle of the scapulae from the stretcher as long as possible until 90 seconds as maximum.
Lower-body flexibility | Patients will be followed over 12 months
  it will be assessed with chair sit and reach test. Patients were instructed to slide their hands as long as possible to touch their toes. The centimeters that were missing (minus score) or exceeded(plus score) from the tip of the foot were registered.

CONTACTS AND LOCATIONS:
Overall Officials: IRENE CANTARERO VILLANUEVA, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Universidad de Granada, Granada, Spain